CLINICAL TRIAL: NCT03030482
Title: Evaluation of Touch Massage on Anxiety in Critically Ill Patients : a Randomised Controlled Trial Study (REaLAX)
Brief Title: Evaluation of Touch Massage on Anxiety in Critically Ill Patients
Acronym: REaLAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Melot Karine, Study principal investigator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P14/10_REaLAX
Record Dates: First submitted 2017-01-21; First posted 2017-01-25 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Anxiety
Keywords: Anxiety; intensive care; mechanical ventilation; touch massage
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Touch massage (Experimental): Patients will have a touch massage session during 30 minutes the intervention will take place remotely (1 h) of all events that can generate anxiety
  Interventions: Procedure: touch massage
- control (No Intervention): standard care ICU

INTERVENTIONS:
Procedure: touch massage — Patients will have a touch massage session during 30 minutes the intervention will take place remotely (1 h) of all events that can generate anxiety
  Arms: Touch massage

SUMMARY:
Anxiety is a common problem encountered in a about 43 % of critically ill patients. Its occurrence can be related to several causes, mainly dominated by invasive procedures.

anxiety management is typically based on a combination of prevention, evaluation, and therapeutic agents. However, it appears important to develop adjuvant approaches. Touch massage is one of them and that has been evaluated in various medical conditions.

The aim of our study is to evaluate the anxiolytic effect of touch massage in critically ill patients during potentially painful nursing procedures.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age≥18 years) hospitalized in Intensive Care Unit > 24 h
* Requiring mechanical ventilation or not
* Securité Sociale affiliated
* Patient with accessible zone for touch massage (head-face, arms-hands, feet, legs and back)
* No significant event (invasive procedure, diagnostic ad, CAT,MRI) before enrollment

Exclusion Criteria:

* Pregnant
* Legal guardianship
* Neurological failure : stroke ischemic or hemorrhagic, meningitis, status epilepticus,polytrauma( including head trauma),meningo encephalitis, meningism,
* Patient with upper limbs neuromuscular disorders
* Cutaneous lesion (zone of touch massage)
* Temperature ≥ 38,5°C
* A positive score of CAM ICU scale
* Patient refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Measure the anxiolytic value of touch massage to critically ill patient, awake, communicating | 60 minutes
  Total score variation of the Spielberger STAI Y-A anxiety scale (short form) before and after the touch massage session (score 6-24) or standard care ICU.

SECONDARY OUTCOMES:
Measure the correlation between the Spielberger STAI Y-A (short form) anxiety scale and the Anxiety Visual Anxiety Scale (EVA-A). | 60 minutes
  Patient anxiety will be evaluated by the score of anxiety measured in millimeters from 0 to 100 using a Visual analogue scale of anxiety (EVA - A) before and after touch massage session or standard care ICU.
Measure the analgesic effect of touch massage to critically ill patient awake, communicating | 60 minutes
  Pain will be evaluated by the pain score measured in millimeters of 0 and 100 with scale visual analog pain (EVA) before and touch massage session or standard care ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Versailles Hospital, Le Chesnay, Yvelines, France

IPD SHARING:
Plan to Share IPD: No